CLINICAL TRIAL: NCT04756752
Title: Effect of a Strength, Endurance and Sports-oriented Rehabilitation Protocol on Functional Mobility and Daily Activity in People With a Lower-limb Amputation
Brief Title: Effect of Sports-oriented Rehabilitation on Mobility and Daily Activity in People With a Lower-limb Amputation
Status: Completed | Type: Observational
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Other Study IDs: 876_Amputatie Parateam
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Amputation; Lower Limb Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fit and Vitaal program: People with a lower-limb amputation participating in the Fit and Vitaal rehabilitation program
  Interventions: Other: Fit and Vitaal program

INTERVENTIONS:
Other: Fit and Vitaal program — Intervention type: training

SUMMARY:
Mobility is one of the most important factors in the quality of life of people with a lower-limb amputation. However, mobility and physical activity are often limited. 61% of amputees is not sufficiently active in daily life and only about 15% of the Dutch amputees regularly participates in sports. Physical inactivity is known to increase the risk of comorbidities, especially among amputation patients who already have a higher prevalence of vascular diseases, diabetes and osteoarthritis. It is clear that sufficient daily physical activity is important to optimize the health and quality of life of amputees.

Research has shown that higher aerobic capacity, higher muscle force and the absence of comorbidities are related to better walking ability, as walking is more energy consuming for people with an amputation. It is therefore expected that increasing strength and cardiovascular fitness results in better mobility, higher daily activity, better physical health and a better quality of life among amputees. To improve physical capacity and sports participation in people with a lower-limb amputation, the Sint Maartenskliniek (Nijmegen, The Netherlands) and Dutch football club N.E.C. Nijmegen developed a new exercise program: Fit en Vitaal. Participants perform a six-week training program with three training sessions each week (fitness, aqua-fitness and a sports and play session) under the guidance of movement agogue. Thereafter, they continue with a low-frequency movement intervention during which they attend various sports clinics once a week for eight months. As social support and contact with peers are important factors in sports participation for amputees, the Fit en Vitaal program was designed as a yearly returning program with a fixed group of participants at the start of each year.

This exploratory study aimed to evaluate both the direct and indirect effects of the Fit en Vitaal program on people with a lower-limb amputation in terms of walking ability, functional mobility, oxygen consumption during walking, daily physical activity at home and experienced quality of life. It is expected that all will improve after the first six weeks of training, and the effects will remain after the eight-month low-frequency training.

DETAILED DESCRIPTION:
Mobility is one of the most important factors in the quality of life of people with a lower-limb amputation.However, many experience limited mobility and show less daily activity compared to healthy individuals. 61% of amputees does not reach a level of sufficiently active in daily life and only about 15% of the Dutch amputees regularly participates in sports. Physical inactivity is known to increase the risk of comorbidities, especially among amputation patients who already have a higher prevalence of vascular diseases, diabetes and osteoarthritis. It is clear that sufficient daily physical activity is important to optimize the health and quality of life of amputees.

A simple way of increasing activity in amputees is increasing their standing and walking duration during the day. Walking is known to require more energy in amputees than in healthy individuals due to their lack of active function in their prosthetic leg. Higher aerobic capacity, higher muscle force and the absence of comorbidities in amputees were already related to better walking ability. Therefore, increasing strength and cardiovascular fitness would presumably result in higher daily activity, physical health and quality of life among amputees.

To improve physical capacity and sports participation in people with a lower-limb amputation, the Sint Maartenskliniek (Nijmegen, The Netherlands) and Dutch football club N.E.C. Nijmegen developed a new exercise program: Fit en Vitaal. Participants perform a six-week training program with three training sessions each week (fitness, aqua-fitness and a sports and play session) under the guidance of movement agogue. Thereafter, they continue with a low-frequency movement intervention during which they attend various sports clinics once a week for eight months. As social support and contact with peers are important factors in sports participation for amputees, the Fit en Vitaal program was designed as a yearly returning program with a fixed group of participants at the start of each year.

This exploratory study aims to evaluate both the direct and indirect effects of the Fit en Vitaal program on people with a lower-limb amputation. Therefore, the primary objective is to evaluate the effect of the program on walking ability, functional mobility and oxygen consumption during walking. As a secondary objective, the effect on daily physical activity at home and experienced quality of life is examined. It is expected that all will improve after the first six weeks of training, and the effect will remain after finishing the eight-month low-frequency training.

ELIGIBILITY:
Inclusion Criteria:

* participation in the Fit en Vitaal program

Exclusion Criteria:

* inability to stand and walk indoors before the start of the study
* other physical therapy or sports participation during the Fit en Vitaal program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a unilateral or bilateral lower-limb amputation participating in the Fit and Vitaal rehabilitation program at the Sint Maartenskliniek, Nijmegen, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
2 Minute Walk Test | 2 minutes
  Measure for walking ability
L-test | 2 minutes
  Measure for functional mobility
Four Square Step Test (FSST) | 2 minutes
  Measure for precision stepping. Highest score: 47. Lowest score: 0.
Amputation Mobility Predictor with prosthesis (AMPPRO) | 15 minutes
  Measure of ambulatory potential
Minutes walking and standing per day | 5 days
  Measure of daily activity, measured with wearable activity sensor
Rand-36 questionnaire | 10 minutes
  Measure of quality of life with 8 domains. Highest score: 100. Lowest score: 0.
VO2/kg/ml | 10 minutes
  Measure of oxygen consumption during walking

CONTACTS AND LOCATIONS:
Overall Officials: Noël LW Keijsers, PhD, Study Chair — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No